CLINICAL TRIAL: NCT06268301
Title: A Randomized, Open-Label, Single-Dose, Two-Way Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics, Safety, and Tolerability of Budesonide Oral Suspension in Healthy Adult Participants
Brief Title: A Study to Determine the Effect Food Has on TAK-721 (Budesonide Oral Suspension) in the Body of Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-721-1003
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: BOS 2 mg Fasted, then Fed (Experimental): Participants will receive 2 mg BOS, single dose, orally on Day 1 of Period 1 under fasted condition (Treatment A). Two days later, participants will receive 2 mg BOS single dose, orally on Day 1 of Period 2 under fed condition (Treatment B).
  Interventions: Drug: Budesonide
- Sequence 2: BOS 2 mg Fed, then Fasted (Experimental): Participants will receive 2 mg BOS, single dose, orally on Day 1 of Period 1 under fed condition (Treatment B). Two days later, participants will receive 2 mg BOS single dose, orally on Day 1 of Period 2 under fasted condition (Treatment A).
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Budesonide oral suspension
  Other Names: TAK-721

SUMMARY:
The main aim of this study is to check what the body of a healthy adult who either fasted or had eaten does to TAK-721 and how TAK-721 is distributed in and removed from the body. Other aims are to learn how safe the treatment with TAK-721 is and how suitable the TAK-721 is for healthy adults who either fasted or had eaten. All participants will receive TAK-721 but half will be assigned by chance to the participant group who are fasting first then getting the high-fat/high-calorie meal later or the group who gets meal first and fasts later. The group assignment will be switched once during the course of the study so that all participants will receive TAK-721 in both a fasted or fed condition.

DETAILED DESCRIPTION:
The drug being tested in this study is called budesonide. Budesonide oral suspension (BOS) is being tested in healthy adult participants. This study will determine whether the absorption of BOS will be altered if taken with food.

The study will enroll approximately 20 patients. The study will consist of two treatment sequences and two periods separated by a washout period of 2 days. Participants will be randomly assigned (by chance, like flipping a fair coin) to one of the two treatment sequences:

* Treatment Sequence 1: Participants will receive 2 mg BOS orally on Day 1 of Period 1 in fasted condition (Treatment A). Two days later, participants will receive 2 mg BOS orally on Day 1 of Period 2 in fed condition (Treatment B).
* Treatment Sequence 2: Participants will receive 2 mg BOS orally on Day 1 of Period 1 in fed condition (Treatment B). Two days later, participants will receive 2 mg BOS orally on Day 1 of Period 2 in fasted condition (Treatment A).

This single center trial will be conducted in the United States. Participation in the study is up to approximately 34 days. Participants will visit the clinic approximately three days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on participant self-reporting.
2. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meters squared (kg/m^2) at the screening visit.

Exclusion Criteria:

1. Presence of any active infection at the screening visit or check-in.
2. Positive urine drug or alcohol results at the screening visit or check-in.
3. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at the screening visit.
4. Participant is unable to refrain from or anticipates the use of:

   1. Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing. Medication listed as part of acceptable birth control methods, hormone replacement therapy, and thyroid hormone replacement medication will be allowed.
   2. Any drugs known to be moderate or strong inducers of cytochrome P450 (CYP) 3A4 enzymes and/or p-glycoprotein (P-gp), including St. John's Wort, for 28 days prior to the first dosing. Appropriate sources (e.g., Flockhart Table™) will be consulted to confirm lack of pharmacokinetic (PK) /pharmacodynamic interaction with the study drug.
5. Participant is lactose intolerant.
6. Donation of blood or significant blood loss within 56 days prior to the first dosing.
7. Plasma donation within 7 days prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/f9368174b21c4a03?idFilter=%5B%22TAK-721-1003%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 6 February 2023 to 20 February 2023.
Pre-assignment Details: Healthy participants were enrolled to receive budesonide oral suspension (BOS) in either of the 2 treatment sequences Fasted-Fed or Fed-Fasted.
Groups:
- Sequence 1: BOS 2 mg Fasted, Then Fed: Participants received 2 mg BOS, single dose, orally on Day 1 of Period 1 under fasted condition (Treatment A). After a washout of at least 2 days participants then received 2 mg BOS single dose, orally on Day 1 of Period 2 under fed condition (Treatment B).
- Sequence 2: BOS 2 mg Fed, Then Fasted: Participants received 2 mg BOS, single dose, orally on Day 1 of Period 1 under fed condition (Treatment B). After a washout of at least 2 days participants received 2 mg BOS single dose, orally on Day 1 of Period 2 under fasted condition (Treatment A).
Period: Period 1
Arm/Group | Sequence 1: BOS 2 mg Fasted, Then Fed | Sequence 2: BOS 2 mg Fed, Then Fasted
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence 1: BOS 2 mg Fasted, Then Fed | Sequence 2: BOS 2 mg Fed, Then Fasted
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: BOS 2 mg Fasted, Then Fed | Sequence 2: BOS 2 mg Fed, Then Fasted | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (9.50) | 32.7 (9.97) | 35.7 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 5 | 6 | 11
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per metre square (kg/m^2)] — BMI = weight (kg)/[height (m)^2]
  kilograms per metre square (kg/m^2) | 27.52 (2.910) | 27.59 (2.706) | 27.56 (2.735)
Height [Mean (Standard Deviation); unit: centimetres (cm)] | 165.4 (10.71) | 169.0 (11.52) | 167.2 (10.98)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 75.99 (15.39) | 79.51 (14.53) | 77.75 (14.68)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: Pharmacokinetic (PK) Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Groups:
- Treatment A: BOS 2 mg Fasted: Participants received 2 mg BOS, single dose, orally on Day 1 of Period 1 or Period 2 under fasted condition.
- Treatment B: BOS 2 mg Fed: Participants received 2 mg BOS, single dose, orally on Day 1 of Period 1 or Period 2 under fed condition.
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
picograms per milliliter (pg/mL) | 692.9 (54.4) | 604.1 (46.6)

2. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms*hours per milliliter (pg*h/mL)
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
picograms*hours per milliliter (pg*h/mL) | 2811 (57.5) | 3529 (52.1)

3. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC∞) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
pg*h/mL | 3075 (57.0) | 3892 (47.1)

4. Secondary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE), Serious Adverse Events (SAE), and Death
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an adverse event with an onset that occurs after receiving study drug. An SAE was defined as any untoward medical occurrence that at any dose results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event that may require an intervention to prevent above items and expose the participant to danger.
Time Frame: From first dose of study drug up to the end of study (EOS) (Up to 15 days)
Population: Safety Set included all participants who received any study drug. Data is presented per fed or fasted condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
Participants
  TEAEs | 2 | 5
  SAEs | 0 | 0
  Deaths | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Sign Values Reported as Adverse Events
Description: Vital signs included body temperature, respiratory rate, blood pressure, and pulse rate evaluations.
Time Frame: From first dose of study drug up to EOS (Up to 15 days)
Population: Safety Set included all participants who received any study drug. Data is presented per fed or fasted condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Clinical Laboratory Values Reported as Adverse Events
Description: Clinical laboratory parameters included hematology, clinical chemistry, serum immunoglobulin and urinalysis tests.
Time Frame: From first dose of study drug up to EOS (Up to 15 days)
Population: Safety Set included all participants who received any study drug. Data is presented per fed or fasted condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

7. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 12 Hours (AUC0-12) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 12 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
pg*h/mL | 2728 (53.0) | 3208 (42.2)

8. Secondary Outcome: Area Under the Curve From the Last Quantifiable Concentration to Infinity Expressed as a Percentage of AUC∞ (AUCextrap%) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
percentage of AUC | 7.275 (61.7) | 7.126 (75.6)

9. Secondary Outcome: Time to First Occurrence of Cmax (Tmax) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
hours (h) | 1.286 [0.55 to 2.57] | 2.516 [1.01 to 6.03]

10. Secondary Outcome: Lag Time to First Quantifiable Concentration (Tlag) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
hours | 0.328 [0.26 to 0.56] | 0.308 [0.25 to 0.53]

11. Secondary Outcome: Terminal Disposition Phase Half-life (t1/2z) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
hours | 4.270 [2.13 to 6.98] | 5.096 [2.78 to 7.35]

12. Secondary Outcome: Terminal Disposition Phase Rate Constant (λz) of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Median (Full Range); unit: 1/hour
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
1/hour | 0.1627 [0.0994 to 0.325] | 0.1362 [0.0943 to 0.249]

13. Secondary Outcome: Apparent Clearance (CL/F) of BOS Calculated Using the Observed Value of the Last Quantifiable Concentration of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
liters per hour (L/h) | 650.4 (57.0) | 513.9 (47.1)

14. Secondary Outcome: Apparent Volume of Distribution During the Terminal Disposition Phase (Vz/F) of BOS Calculated Using the Observed Value of the Last Quantifiable Concentration of BOS
Time Frame: Periods 1 and 2: Pre-dose and at multiple timepoints (up to 24 hours) post-dose on Day 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
Number analyzed (Participants) | 20 | 20
liters (L) | 3967 (45.0) | 3513 (32.9)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to the EOS (15 days)
Description: Safety Set included all participants who received any study drug. Data is presented per fed or fasted condition.
Arm/Group | Treatment A: BOS 2 mg Fasted | Treatment B: BOS 2 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: BOS 2 mg Fasted (N=20) | Treatment B: BOS 2 mg Fed (N=20)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 2
Vessel puncture site bruise (General disorders) | 0 | 1
Vessel puncture site swelling (General disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT06268301/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT06268301/SAP_001.pdf